CLINICAL TRIAL: NCT01126840
Title: Cancer Survivorship in Lynch Syndrome: Impact on Patients and Families
Brief Title: Survivorship in Lynch Syndrome Families
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2010-0160; CA57730 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer
Keywords: Lynch Syndrome; Families; Quality of life; QOL; First-degree relatives; Questionnaire; Interview
MeSH Terms: conditions — Colorectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire + Telephone Interview: Mailed questionnaire that contains questions about experiences living with colorectal cancer, take 45-60 minutes to complete. The phone interview should take 30-45 minutes to complete.
  Interventions: Behavioral: Telephone Interview; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Telephone Interview — The phone interview should take 30-45 minutes to complete.
  Other Names: Survey
Behavioral: Questionnaire — Mailed questionnaire that contains questions about experiences living with colorectal cancer, take 45-60 minutes to complete.
  Other Names: Survey

SUMMARY:
Objectives:

Specific Aims:

1. Researchers will evaluate and compare predictors of health-related quality of life (QOL) among colorectal cancer (CRC) survivors who have Lynch syndrome (LS) with those patients who have sporadic CRC using both quantitative and qualitative methodology.

   a. In both CRC groups, researchers will evaluate cancer preventive and health behaviors, including lifestyle factors and screening, psychosocial factors, including mood, family functioning, coping style, anxiety, depression, and social resources, and health care system factors, including interactions with health care providers and service utilization.
2. Researchers will compare the experience of first-degree relatives (FDRs) of patients who have LS with that of FDRs of patients who have sporadic CRC using both quantitative and qualitative methodology.

   a. Researchers will evaluate all of the domains listed above, as well as anticipatory grief, assessment of caregiving responsibilities, and fear of cancer in FDRs of patients with LS-related and sporadic CRC.
3. Researchers will examine CRC patients from both groups and their FDRs using dyadic analyses in order to evaluate the similarities and differences in their survivorship experience.
4. Researchers will evaluate the preventive and health behavior of patients who are non-conclusive for Lynch syndrome and their family members. They will examine their screening behavior and will explore how the interaction between the patients and their relatives affects the relatives' screening behavior. They also will examine how these non conclusive LS patients and their family members perceive their risk for LS-related cancers.

DETAILED DESCRIPTION:
Data will be collected primarily using a mailed self-administered questionnaire. A subset of the participants who complete the mailed questionnaire will be recontacted and invited to participate in an in-depth, semi-structured telephone interview.

Qualitative Mailed Questionnaires:

Participants will complete a questionnaire that contains questions about your experiences living with colorectal cancer. The questionnaire should take 45-60 minutes to complete.

Up to 200 colorectal cancer survivors and up to 200 close relatives of colorectal cancer survivors will take part in this portion of the study.

Telephone Interviews:

In the phone interview, you will be asked some questions about your experiences living with colorectal cancer. The phone interview should take 30-45 minutes to complete.

Up to 30 colorectal cancer survivors and up to 30 close relatives of colorectal cancer survivors will take part in this portion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal cancer (CRC) patients with Lynch-syndrome related CRC: Diagnosis of CRC
2. Colorectal cancer (CRC) patients with sporadic CRC: Diagnosis of CRC
3. All First-degree relatives (FDRs): Siblings or adult children of recruited CRC patients
4. All Participants: 18 years of age or older
5. All Participants: Able to read and speak English
6. All Participants: Able to be contacted by mail.
7. All Second and Third relatives (SDRs and TDRs): Grandparents, grandchildren, aunts, uncles, nieces, nephews, and first-degree cousins of recruited CRC patients
8. IPs with a LS MMR mutation who were seen at MDACC for genetic counseling and testing during 2011-2014.

Exclusion Criteria:

1) CRC patients with sporadic CRC: Personal or family history of Lynch syndrome, familial adenomatous polyposis, inflammatory bowel disease or those who have a FDR with CRC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer (CRC) patients with Lynch-syndrome related CRC or with sporadic CRC; along with first-degree relatives (FDRs), Siblings or adult children of recruited CRC patients
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2010-06-20 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Compare Predictors of Health-Related Quality of Life (QOL) among Colorectal Cancer (CRC) Survivors who have Lynch Syndrome (LS) with patients who have Sporadic CRC | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, MPH,PHD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org